CLINICAL TRIAL: NCT07205419
Title: Application of an Eye-Tracking Interaction System for Non-verbal ICU Patients Based on Co-Design Principles: A Feasibility Randomized Controlled Trial With an Embedded Qualitative Study
Brief Title: Eye-Tracking Interaction System for Non-verbal ICU Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ZS202500100
Record Dates: First submitted 2025-09-02; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Communication Barriers; Eye-tracking Technology; ICU Patients

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group: (No Intervention): Charge nurses will lead communication through body language (e.g., pointing, nodding, shaking the head) or by providing writing boards for patients to write. Patients unable to write will communicate solely through body language.
- Intervention Group (Experimental): Charge nurses will lead communication using the eye-tracking interaction system. An eye-tracking interaction system refers to an eye-tracking interaction interface installed on any electronic device equipped with a camera that meets the configuration requirements.
  Interventions: Device: Eye-Tracking Interaction System

INTERVENTIONS:
Device: Eye-Tracking Interaction System — The eye-tracking interactive interface designed based on evidence-based and co-design principles is installed on tablets or computers equipped with cameras, forming the eye-tracking interactive system.
  Arms: Intervention Group

SUMMARY:
The objectives of this clinical trial are to explore the feasibility of the eye-tracking interactive system in improving communication disorders among non-verbal ICU patients. It will also preliminarily investigate the effectiveness of this system in facilitating communication for these patients.

Researchers will compare the eye-tracking interactive system with traditional augmentative and alternative communication (AAC) technologies (such as body language, writing boards, etc.) to observe the feasibility and preliminary effectiveness of the eye-tracking interactive system in improving communication disorders.

Participants will:

* Use augmentative and alternative communication technologies daily
* Have detailed records of every communication interaction

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Patients in the ICU who are unable to communicate through normal verbal means due to endotracheal intubation/tracheotomy, muscle or nerve injury, acute/chronic spinal cord injury, etc.
* Richmond Agitation-Sedation Scale (RASS) score of -1 to 1;④Primary caregivers are adults
* Able to read Chinese characters and follow simple commands
* Willing to participate in this study

Exclusion Criteria:

* Diseases associated with cognitive impairment, such as pulmonary encephalopathy, hepatic encephalopathy, diabetic hyperosmolar coma, and coma of unknown cause
* A history of mental disorders, dementia or pre-dementia, or intellectual disability
* Conditions precluding cooperation with eye-tracking interaction, such as blindness or inability to elevate the eyelids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Communication efficiency | up to 5 days after enrollment
  Communication efficiency is defined as the number of correctly expressed needs per minute, calculated as the total number of correctly expressed needs divided by the duration in minutes. The aforementioned duration of assistive communication and total number of correctly expressed needs will be documented in the Communication Information Registration Form.
Communication accuracy | up to 5 days after enrollment
  Communication accuracy is calculated as the number of correctly expressed needs divided by the total number of expressed needs. The aforementioned total number of expressed needs and total number of correctly expressed needs will be documented in the Communication Information Registration Form.
Patients' communication ability | up to 5 days after enrollment
  The LCS (Loewenstein Communication Scale) will be used to assess patients' communication ability. This tool is primarily used in clinical practice to assess the communication abilities of minimally responsive patients. It comprises five hierarchical functions: mobility, respiration, visual responsiveness, auditory comprehension, and communication. Each function is divided into five parameters, with scores ranging from 0 to 4 (each function has a maximum score of 20, and the total score is 100).

SECONDARY OUTCOMES:
Nurses' compliance | through study completion, an average of 1 year
  The compliance of nurses is defined as the number of times nurses in the intervention group use the eye-tracking interactive system for assistive communication divided by the total number of communication interactions.
Time spent training patients during initial use | Day 1
  The research team is going to independently develop a Communication Information Registration Form, which is to include the duration of training provided by nurses to patients when they use the eye-tracking interactive system for the first time. After the completion of the intervention, the average training duration is to be calculated.
Incidence of delirium | at 9:00 AM and 9:00 PM daily
  The CAM-ICU (Confusion Assessment Method for the Intensive Care Unit) will be used to assess the occurrence of delirium.The CAM-ICU uses the CAM algorithm and has four features: (1) altered mental status/fluctuating course, (2) inattention, (3) altered level of consciousness, and (4) disorganized thinking. Like the CAM, a patient must be inattentive (cardinal feature of delirium) in order to be CAM-ICU positive.
Patient satisfaction | up to 5 days after enrollment
  The PIADS (Psychosocial Impact of Assistive Devices Scale) will be used to measure the impact of assistive devices on patients and their satisfaction levels.This tool is a 26-item, self-report questionnaire designed to assess the effects of an assistive device on functional independence, well-being, and quality of life. Each item is rated on a 7-point Likert scale, ranging from -3 to +3. Higher scores generally indicate that the assistive device has a more positive impact on these aspects; conversely, lower scores suggest a less positive impact, or even potential negative effects.
Patient enrollment rate | through study completion, an average of 1 year
  The patient enrollment rate is calculated as the number of patients who successfully meet the eligibility criteria and are enrolled in the study divided by the total number of patients screened for eligibility during the study period.
Patient withdrawal rate | through study completion, an average of 1 year
  The patient withdrawal rate is defined as the number of enrolled patients who discontinue study participation (for any reason) prior to the completion of the predefined study protocol (e.g., intervention course) divided by the total number of enrolled patients.